CLINICAL TRIAL: NCT05432102
Title: Patient Experience and Technical Success of Community Sleep Studies
Acronym: PETSOCSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Iceni Laboratories (Unknown); CRN Eastern (Unknown)
Responsible Party: Sponsor
Other Study IDs: P02530
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants having respiratory polygraphy: This label will used to describe participants having respiratory polygraphy at Royal Papworth Hospital over a 3 month period.
  Interventions: Diagnostic Test: Respiratory polygraphy
- Participants having pulse oximetry: This label will used to describe participants having pulse oximetry at Royal Papworth Hospital over a 3 month period.
  Interventions: Diagnostic Test: Pulse oxymetry

INTERVENTIONS:
Diagnostic Test: Pulse oxymetry — Diagnostic intervention to diagnose OSA.
  Groups: Participants having pulse oximetry
Diagnostic Test: Respiratory polygraphy — Diagnostic intervention to diagnose OSA.
  Groups: Participants having respiratory polygraphy

SUMMARY:
This study looks at the quality of the common mechanisms used to diagnose obstructive sleep apnoea (OSA) by patients in their own homes. These are pulse oximetry as a stand alone measurement and multi-channel respiratory studies that measure oximetry but also record some combination of signals including airflow at the mouth and or nose, chest and abdominal expansion, body position and snoring. This study will examine the patient acceptability of these methods and the proportion of studies that achieve various levels of technical quality ranging from a full night with all data available to a completely failed study and categories in between.

DETAILED DESCRIPTION:
There is a study underway to develop a non-contact detector of breathing (SafeScan) as a new method of diagnosing obstructive sleep apnoea (OSA). There are a number of different methods already available to achieve this end but one proposed advantage of the new SafeScan device is that it will not affect sleep quality and because there are no measuring devices attached to the patient it is less likely that the signal will be lost in the night due to the normal movements of sleep. However there are no data available that quantify these factors as an issue for the current techniques and devices.

The proving study for SafeScan is a comparison of the ability of the device to measure sleep apnoea compared to full in-hospital polysomnography (PSG) and one outcome will be the proportion of studies that have lost data. However the future use of the SafeScan device will be in the community. The common diagnostics used by patients in their own homes are pulse oximetry as a stand alone measurement and multi-channel respiratory studies that measure oximetry but also record some combination of signals including airflow at the mouth and or nose, chest and abdominal expansion, body position and snoring. We propose a study to examine the patient acceptability of these methods and the proportion of studies that achieve various levels of technical quality ranging from a full night with all data available to a completely failed study and categories in between. In addition there will be an analysis of the results to explore whether there are features of the patients such as age and obesity that make technical success or failure of the studies more likely.

ELIGIBILITY:
Inclusion Criteria:

Patient able to provide assent by completion of the Research Questionnaire Adult patients (≥ 18 years of age) Patients undergoing a home sleep study

Exclusion Criteria:

Patients unable to complete questionnaires due to language or other barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a home sleep study at Royal Papworth Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Satisfactory sleep studies | 3 months
  The proportion of home studies to diagnose sleep apnoea that are satisfactory without disruption to the patient's sleep or loss of signals to an extent that make the results unreliable.

SECONDARY OUTCOMES:
Extent of sleep disruption | 3 months
  What proportion of patients report sleep disruption due to: oximeter probe / nasal cannula / thermistor / chest band /abdominal band / the recording device?
Extent of signal failure | 3 months
  What proportion of studies failed due to loss of signal from: oximeter probe / nasal cannula / thermistor / chest band /abdominal band / the recording device?

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, United Kingdom